CLINICAL TRIAL: NCT03081949
Title: Peripartum Cardiomyopathy in Nigeria (PEACE) A Registry to Study the Demographics, Social and Clinical Characteristics, Pathophysiology and Outcomes of Peripartum Cardiomyopathy in Nigeria
Brief Title: Peripartum Cardiomyopathy in Nigeria Registry
Acronym: PEACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aminu Kano Teaching Hospital (Other)
Collaborators: Nigerian Cardiac Society (Unknown)
Responsible Party: Principal Investigator, Prof Kamilu Karaye, Professor and Honorary Consultant, Aminu Kano Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: version 3
Record Dates: First submitted 2017-02-22; First posted 2017-03-17 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Peripartum Cardiomyopathy
Keywords: peripartum cardiomyopathy; Ventricular remodelling; Survival; Selenium; Oxidative stress; Nigeria
MeSH Terms: conditions — Peripartum Cardiomyopathy; Ventricular Remodeling | interventions — Sodium Selenite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Oral Sodium Selenite 200 µg/day for 3 months
  Interventions: Drug: Oral Sodium Selenite 200 µg/day for 3 months
- Control (No Intervention): No treatment

INTERVENTIONS:
Drug: Oral Sodium Selenite 200 µg/day for 3 months — PPCM patients with selenium deficiency, who have not achieved LV reverse remodelling (LVRR) (LV end-diastolic dimension indexed to body surface area (LVEDDi) ≤33.0 mm/m2) at 6 months after diagnosis.
  Other Names: Nature's way Selenium 200mcg
  Arms: Treatment

SUMMARY:
Peripartum cardiomyopathy (PPCM) is a global disease with significant morbidity and mortality, and Nigeria probably has the highest burden of the disease in the world. Unfortunately, much about the disease including its aetiology, epidemiology and treatment is not yet well described. This will be a prospective, national, multicenter cohort study, conducted in centres in Nigeria. It is expected that approximately 500 patients with PPCM and 500 apparently healthy pregnant women will be recruited over a 6-month period with follow-up at 3-monthly intervals for 18 months.

DETAILED DESCRIPTION:
Peripartum cardiomyopathy (PPCM) is a global disease with significant morbidity and mortality, and Nigeria probably has the highest burden of the disease in the world. Unfortunately, much about the disease including its aetiology, epidemiology and treatment is not yet well described. This will be a prospective, national, multicenter cohort study, conducted in centres in Nigeria. It is expected that approximately 500 patients with PPCM and 500 apparently healthy pregnant women will be recruited over a 6-month period with follow-up at 3-monthly intervals for 18 months. The objectives of the study are:

i. To describe the burden and demographic, social and clinical characteristics of PPCM in Nigeria.

ii. To describe the ventricular remodelling and outcomes (rehospitalisation rate, cardio-embolic events and survival) of PPCM in Nigeria.

Sub-study:

iii. To study the relationship between selenium deficiency, oxidative stress and PPCM in Nigeria.

iv. To describe the prevalence of selenium deficiency and its relationship with cardiac function in apparently healthy pregnant women in Nigeria.

v. To study the impact of sodium selenite supplementation on cardiac function among selenium deficient PPCM patients who have not recovered left ventricular function at 6 months after the diagnosis.

This will be the largest systematic evaluation of PPCM in Nigeria, and it is hoped that the information will assist in developing locally applicable treatment guidelines, policies and interventions for this seemingly deadly disease.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PPCM
* PPCM patients with HF symptoms at the time of recruitment
* Asymptomatic pregnant women attending antenatal clinic (ANC)
* Sub-study: Open-label randomised Trial: Non-pregnant PPCM patients with all of the following: LVEF <35% and/or LVEDDi≤33.0 mm/m2 at 6 months postpartum AND selenium deficiency
* Written informed consent

Exclusion Criteria:

* Asymptomatic PPCM patients at the time of recruitment
* PPCM patients who are not expected to survive at least 6 months from recruitment
* Pregnant women with any medical condition other than PPCM
* Subjects who are considered not likely to attend follow up reviews regularly, because of lack of patient's and close relative's phone numbers, or long distance from the study centre, etc
* Refusal or withdrawal of consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of peripartum cardiomyopathy (PPCM) in Nigeria | Over 6 months
  All participants confirmed to have PPCM presenting to the study centres, as described in PEACE Registry protocol V3.

SECONDARY OUTCOMES:
Selenium deficiency in PPCM patients and apparently healthy pregnant women in Nigeria | At baseline, 3 months, 12 and 18 months of follow up.
  Prevalence of selenium deficiency will be assessed. Serum selenium will be measured as described in PEACE Registry protocol V3. Selenium deficiency will be defined as serum selenium <70μg/L.
Oxidative stress in PPCM patients and apparently healthy pregnant women in Nigeria | At baseline, 3 months, 12 and 18 months of follow up.
  Prevalence of oxidative stress will be assessed. Serum malondialdehyde (MDA), superoxide dismutase (SOD), glutathione peroxidise (GPO) and N-terminal pro-B-type natriuretic peptide (NT-BNP) will be measured as described in PEACE Registry protocol V3. Abnormal oxidative stress will be defined as the presence of serum NT-BNP >125pg/mL and ANY of the following: plasma MDA >1.25μmol/L, serum SOD >110ng/mL and plasma GPO >470U/L.
The effect of sodium selenite supplementation on cardiac function among PPCM patients. | 18 months
  PPCM patients with selenium deficiency, left ventricular ejection fraction (LVEF) <35% and/or insignificant left ventricular reverse remodeling (LVRR) at 6 months postpartum, will be offered sodium selenite 200mcg daily for 3 months, in an open-label randomized trial. LVRR would be defined as the presence of both absolute increase in LVEF ≥10.0% and decrease in LV end-diastolic dimension indexed to body surface area (LVEDDi) ≤33.0 mm/m2, while recovered LV systolic function as LVEF ≥55%, during the follow-up.
  Change in LVEF and LVEDDi will be measured at 6, 12, and 18 months follow up visits, to determine prevalence of LVRR among partipants on selenium treatment and those who will not be on selenium treatment.
Left Ventricular remodelling in PPCM patients | At baseline, and 6, 12 and18 months follow up
  Change in LVEF and LVEDDi to determine LVRR
Right Ventricular (RV) remodelling in PPCM patients | At baseline, and 6, 12 and18 months follow up
  Change in RV fractional area change (RVFAC) of the right ventricle (in cm2), to determine RV reverse remodelling (RVRR). RVRR is defined as RVFAC >35cm2.
Rehospitalisation rate | 18 months
  Number of participants who experience hospitalization for any cardiovascular disease during follow up.
Prevalence of cardio-embolic events | 18 months
  Number of participants who experience stroke, transient ischemic attack or any gangrene during the follow-up period of the study.
Survival rate | 18 months
  Number of participants who have survived the follow-up period of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Kamilu M Karaye, PhD, Principal Investigator — Aminu Kano Teaching Hospital, Kano
Locations (1):
- Aminu Kano Teaching Hospital, Kano, Nigeria

IPD SHARING:
Plan to Share IPD: No
We intend to publish the results in peer reviewed scientific journals.

REFERENCES:
- [Result] Karaye KM, Sa'idu H, Balarabe SA, Ishaq NA, Sanni B, Abubakar H, Mohammed BL, Abdulsalam T, Tukur J, Mohammed IY. Selenium supplementation in patients with peripartum cardiomyopathy: a proof-of-concept trial. BMC Cardiovasc Disord. 2020 Oct 21;20(1):457. doi: 10.1186/s12872-020-01739-z. PMID 33087055
- [Result] Karaye KM, Sa'idu H, Balarabe SA, Ishaq NA, Sanni B, Abubakar H, Mohammed BL, Abdulsalam T, Tukur J, Mohammed IY. Correction to: Selenium supplementation in patients with peripartum cardiomyopathy: a proof-of-concept trial. BMC Cardiovasc Disord. 2021 Jan 4;21(1):4. doi: 10.1186/s12872-020-01782-w. No abstract available. PMID 33397290